CLINICAL TRIAL: NCT02648412
Title: Pupillary Diameter Variation After Standardized Tetanic Stimulations of Incremental Intensities in Patients Under Ketamine Sedation
Brief Title: Pupillary Dilation After Incremental Tetanic Stimulations Under Ketamine Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pupillo ketamine
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Pain; Anesthesia
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine sedation (Experimental): Procedure scheduled under ketamine sedation. Baseline pupillary diameter measurement in alert subjects. Injection of a bolus of 1 mg/kg of ketamine. Every minute, tetanic stimulations of incremental intensities (10-20-30-40-60 milliamps), during 5 seconds.
  Pupillary diameter measurement before and after each stimulation. End of study period, beginning of procedure.
  Interventions: Drug: ketamine; Procedure: Tetanic stimulations of incremental intensities

INTERVENTIONS:
Drug: ketamine — bolus 1 mg/kg
Procedure: Tetanic stimulations of incremental intensities — 10-20-30-40-60 milliamps on the patient's left forearm

SUMMARY:
The aim of the study was to describe the relationship between the intensity of a standardized tetanic stimulation and the associated reflex pupillary dilation in patients under ketamine sedation.

After an intravenous bolus of 1 mg/kg of ketamine, tetanic stimulations were performed every minute at increasing intensities of 10, 20, 30, 40 and 60 milliamps (similar to the stimulations of neuromuscular blocking agents monitoring). Pupillary diameter was measured before and after each stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to pediatric burns care unit
* Burnt skin area 5-40%
* Scheduled for a dressing change under ketamine sedation

Exclusion Criteria:

* Neurologic or ophthalmic disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pupillary dilation: difference between post- and pre-stimulation pupillary diameter assessed by videopupillometry | 30 seconds after each stimulation (6 stimulations per patient)
  Non-invasive measurement of pupillary diameter using an infrared camera, for each of the 6 stimulations per patient

SECONDARY OUTCOMES:
Heart rate variation | 30 seconds after each stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, PHD, Study Director — University Hospital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France